CLINICAL TRIAL: NCT05869487
Title: Evaluation of a Diagnostic Method: Calf Circumference Versus X-ray Absorptiometry in the Diagnosis of Sarcopenia in Elderly Hospitalized Participants
Brief Title: Calf Circumference Versus X-ray Absorptiometry in the Diagnosis of Sarcopenia in Elderly Hospitalized Patients
Acronym: PAPY-SARCM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHRO-2023-02
Record Dates: First submitted 2023-05-11; First posted 2023-05-22 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Sarcopenia
Keywords: Sarcopenia; Absorptiometry; Photon
MeSH Terms: conditions — Sarcopenia | interventions — Absorptiometry, Photon

STUDY DESIGN:
Intervention Model Description: This is a prospective single-center evaluation of a diagnostic method
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- X-ray (Other): Whole body x-ray absorptiometry for measurement of appendicular muscle mass in kilograms. Only one measurement per participant.
  Interventions: Radiation: Dual-energy X-ray absorptiometry

INTERVENTIONS:
Radiation: Dual-energy X-ray absorptiometry — Whole body x-ray absorptiometry

SUMMARY:
This is a prospective single-center study to evaluate a diagnostic method. The main objective of the study is to evaluate the performance of calf circumference as a diagnostic method for sarcopenia in hospitalized elderly people, compared to a gold standard method which is X-ray absorptiometry. The study population are hospitalizing participants aged 75 years and older with an indication to search for sarcopenia.

DETAILED DESCRIPTION:
Sarcopenia is a loss of muscle mass associated with a loss of muscle strength. Sarcopenia is associated with an increase of mortality, risk of falling and hospitalization. The gold standard for assessing loss of muscle mass is X-ray absorptiometry. However, this exam is not systematically performed. The calf circumference (cutoff less than 31 centimeters) is preferentially used. However, this cutoff was defined from a population of women with a mean age of 80 years and a unfrail phenotypic profile that does not allow this result to be applied to elderly hospitalized patients.

The main objective of this study is to evaluate the performance of calf circumference as a diagnostic method for sarcopenia in hospitalized elderly people, compared to a gold standard method which is X-ray absorptiometry.

This is a single-center prospective study to evaluate a diagnostic method. The participants in the study will be hospitalized patients aged 75 years and over, with an indication to search for sarcopenia in the context of screening for protein-energy undernutrition under the recommendations of the French National Authority for Health. Participants will be included after being informed about the protocol and after obtaining their free and informed oral consent. Measurement of calf circumference will be performed before absorptiometry, the results of which will be analyzed in a blinded. The number of subjects to be included with a expected prevalence of 75%, specificity of 95% and an accuracy of 2% is 298 participants according to the literature. A sensitivity and specificity analysis will be performed using the ROC curve. A linear regression analysis will be performed with a significance threshold for the alpha risk of 5%.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 75 years
* Hospitalization in a medical department or in the follow-up care or rehabilitation department of the Hospital Center of Orléans
* Presence of an etiological criterion of undernutrition
* Presence of a decrease in muscle strength

Exclusion Criteria:

* Presence of one of two phenotypic criteria for undernutrition other than sarcopenia, which are body mass index less than 22 kilogram per square meter and weight loss (≥ 5 percent over 1 month or ≥ 10 percent over 6 months or ≥10 percent compared with usual weight before the disease).
* Refusal to participate in the study
* Patient under legal protection
* Impossible to perform X-ray absorptiometry (behavioral problems, functional constraints to climb on the DXA machine)
* Person not affiliated to a social security system

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 298 (Estimated)
Dates: Start 2023-12-11 (Actual); Primary Completion 2027-04-11 (Estimated); Study Completion 2027-04-11 (Estimated)

PRIMARY OUTCOMES:
Measurement of muscle mass using calf circumference | Day 2
  Measurement with a tape measure (in centimetres) of the maximum circumference of the calf
Measurement of muscle mass using X-ray absorptiometry | Day 2
  Measurement of appendicular mass by X-ray absorptiometry in kilograms

SECONDARY OUTCOMES:
Arm circumference | Day 0
  Measurement with a tape measure (in centimetres) of the maximum circumference of the arm
Circumference of the thigh | Day 0
  Measurement with a tape measure (in centimetres) of the maximum circumference of the thigh

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu COULONGEAT, MD, Principal Investigator — CHR d'Orléans
Locations (1):
- CHU d'Orléans, Orléans, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Librero J, Peiro S, Ordinana R. Chronic comorbidity and outcomes of hospital care: length of stay, mortality, and readmission at 30 and 365 days. J Clin Epidemiol. 1999 Mar;52(3):171-9. doi: 10.1016/s0895-4356(98)00160-7. PMID 10210233
- [Result] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jan 1;48(1):16-31. doi: 10.1093/ageing/afy169. PMID 30312372
- [Result] Rolland Y, Lauwers-Cances V, Cournot M, Nourhashemi F, Reynish W, Riviere D, Vellas B, Grandjean H. Sarcopenia, calf circumference, and physical function of elderly women: a cross-sectional study. J Am Geriatr Soc. 2003 Aug;51(8):1120-4. doi: 10.1046/j.1532-5415.2003.51362.x. PMID 12890076
- [Result] Beaudart C, Zaaria M, Pasleau F, Reginster JY, Bruyere O. Health Outcomes of Sarcopenia: A Systematic Review and Meta-Analysis. PLoS One. 2017 Jan 17;12(1):e0169548. doi: 10.1371/journal.pone.0169548. eCollection 2017. PMID 28095426
- [Result] Pagotto V, Santos KFD, Malaquias SG, Bachion MM, Silveira EA. Calf circumference: clinical validation for evaluation of muscle mass in the elderly. Rev Bras Enferm. 2018 Mar-Apr;71(2):322-328. doi: 10.1590/0034-7167-2017-0121. English, Portuguese. PMID 29412289
- [Result] Kawakami R, Murakami H, Sanada K, Tanaka N, Sawada SS, Tabata I, Higuchi M, Miyachi M. Calf circumference as a surrogate marker of muscle mass for diagnosing sarcopenia in Japanese men and women. Geriatr Gerontol Int. 2015 Aug;15(8):969-76. doi: 10.1111/ggi.12377. Epub 2014 Sep 20. PMID 25243821
- [Result] Bahat G, Tufan A, Tufan F, Kilic C, Akpinar TS, Kose M, Erten N, Karan MA, Cruz-Jentoft AJ. Cut-off points to identify sarcopenia according to European Working Group on Sarcopenia in Older People (EWGSOP) definition. Clin Nutr. 2016 Dec;35(6):1557-1563. doi: 10.1016/j.clnu.2016.02.002. Epub 2016 Feb 11. PMID 26922142
- [Result] Maeda K, Koga T, Nasu T, Takaki M, Akagi J. Predictive Accuracy of Calf Circumference Measurements to Detect Decreased Skeletal Muscle Mass and European Society for Clinical Nutrition and Metabolism-Defined Malnutrition in Hospitalized Older Patients. Ann Nutr Metab. 2017;71(1-2):10-15. doi: 10.1159/000478707. Epub 2017 Jun 24. PMID 28647743
- [Result] Roberts HC, Denison HJ, Martin HJ, Patel HP, Syddall H, Cooper C, Sayer AA. A review of the measurement of grip strength in clinical and epidemiological studies: towards a standardised approach. Age Ageing. 2011 Jul;40(4):423-9. doi: 10.1093/ageing/afr051. Epub 2011 May 30. PMID 21624928
- [Result] Dodds RM, Syddall HE, Cooper R, Benzeval M, Deary IJ, Dennison EM, Der G, Gale CR, Inskip HM, Jagger C, Kirkwood TB, Lawlor DA, Robinson SM, Starr JM, Steptoe A, Tilling K, Kuh D, Cooper C, Sayer AA. Grip strength across the life course: normative data from twelve British studies. PLoS One. 2014 Dec 4;9(12):e113637. doi: 10.1371/journal.pone.0113637. eCollection 2014. PMID 25474696
- [Result] Studenski SA, Peters KW, Alley DE, Cawthon PM, McLean RR, Harris TB, Ferrucci L, Guralnik JM, Fragala MS, Kenny AM, Kiel DP, Kritchevsky SB, Shardell MD, Dam TT, Vassileva MT. The FNIH sarcopenia project: rationale, study description, conference recommendations, and final estimates. J Gerontol A Biol Sci Med Sci. 2014 May;69(5):547-58. doi: 10.1093/gerona/glu010. PMID 24737557
- [Result] Gould H, Brennan SL, Kotowicz MA, Nicholson GC, Pasco JA. Total and appendicular lean mass reference ranges for Australian men and women: the Geelong osteoporosis study. Calcif Tissue Int. 2014 Apr;94(4):363-72. doi: 10.1007/s00223-013-9830-7. Epub 2014 Jan 5. PMID 24390582
- [Result] Cheng KY, Chow SK, Hung VW, Wong CH, Wong RM, Tsang CS, Kwok T, Cheung WH. Diagnosis of sarcopenia by evaluating skeletal muscle mass by adjusted bioimpedance analysis validated with dual-energy X-ray absorptiometry. J Cachexia Sarcopenia Muscle. 2021 Dec;12(6):2163-2173. doi: 10.1002/jcsm.12825. Epub 2021 Oct 4. PMID 34609065